CLINICAL TRIAL: NCT00755781
Title: A Multi-Center, Randomized, Controlled Study to Demonstrate the Efficacy and Safety of Cyclosporine Inhalation Solution (CIS) in Improving Bronchiolitis Obliterans Syndrome-Free Survival Following Lung Transplantation
Brief Title: Study of Cyclosporine Inhalation Solution (CIS) in Improving Bronchiolitis Obliterans Syndrome-Free Survival Following Lung Transplantation
Acronym: CIS001
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: APT Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CIS001
Record Dates: First submitted 2008-09-17; First posted 2008-09-19 (Estimated); Last update posted 2012-09-17 (Estimated); Status verified 2012-09

CONDITIONS: Lung Transplant
Keywords: lung transplant; lung transplant recipient; bronchiolitis obliterans syndrome; bronchiolitis obliterans; single lung transplant; double lung transplant; heart-lung transplant; Aerosol
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome; Bronchiolitis Obliterans | interventions — Cyclosporine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CIS (Active Comparator): CIS in addition to standard immunosuppressive regimen.
  Interventions: Drug: Cyclosporine Inhalation Solution (CIS)
- SOC (No Intervention): Standard of care (SOC) therapy for lung transplant recipients

INTERVENTIONS:
Drug: Cyclosporine Inhalation Solution (CIS) — Cyclosporine (USP) Inhalation Solution; 300mg/4.8 mL in propylene glycol (USP) at a concentration of 62.5 mg/mL; 3 times a week for study duration (up to 3 years)
  Other Names: Cyclosporine
  Arms: CIS

SUMMARY:
A Phase III, multi-center, randomized, controlled study designed to demonstrate the efficacy and safety of Cyclosporine Inhalation Solution (CIS)in improving survival and preventing bronchiolitis obliterans syndrome (BOS) when given prophylactically to lung transplant recipients in addition to their standard immunosuppressive regimen.

ELIGIBILITY:
Inclusion Criteria:

* A recipient of a single or double lung transplant (including heart-lung transplant)
* Age 18 years or older
* Able to produce a forced expiratory volume in one second (FEV1) of greater than one liter at randomization
* Eligible subjects must be enrolled within 70 days after receiving a lung transplant
* Clinical status sufficiently stable to enable routine post-transplant bronchoscopy with bronchoalveolar lavage (BAL) and chest X-ray (or equivalent i.e., chest computerized tomogram (CT)) prior to screening

Exclusion Criteria:

* Lung re-transplantation
* Documented allergy to propylene glycol and/or cyclosporine
* Documented respiratory or anastomotic infections unless on appropriate antimicrobial therapy with evidence of clinical response
* Women who are pregnant, wishing to become pregnant, or unwilling to use appropriate birth control to avoid becoming pregnant
* Women who are breastfeeding
* Clinically significant bronchial stenosis unresponsive to dilation and/or stenting
* Malignancies diagnosed within one year prior to screening (with the exception of non-melanomatous skin cancers)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 284 (Actual)
Dates: Start 2008-09; Primary Completion 2011-09 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Duration of BOS-free survival. Other causes for the decline should be excluded by bronchoscopy and other diagnostic testing performed at the discretion of the investigator. The diagnosis of BOS will be determined by the Outcomes Committee | Assessed when symptoms of syndrome present

SECONDARY OUTCOMES:
Pulmonary function as measured by mean FEV1 percent predicted at 2 years after randomization | From study initiation through 2+ years after randomization
All cause mortality | From study initiation through 2+ years after randomization
Duration of event-free survival, corresponding to the length of time between date of randomization and either death or the occurrence of serious bacterial and viral infections that start in the lungs (defined by reporting of a SAE) | From study initiation through 2+ year after randomzation

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Dilly, MD PhD, Study Director — APT Pharmaceuticals, Inc.
Locations (19):
- United States (18):
  - UCLA School of Medicine, Los Angeles, California
  - University of California, San Francisco, San Francisco, California
  - Stanford University Medical Center, Stanford, California
  - University of Colorado Health Sciences Center, Denver, Colorado
  - University of Florida Health Sciences Center, Gainesville, Florida
  - Mayo Clinic, Jacksonville, Florida
  - Tampa General Hospital, Tampa, Florida
  - University of Chicago Hospitals, Chicago, Illinois
  - Loyola University Hospital, Maywood, Illinois
  - Indiana Methodist Research Institute, Indianapolis, Indiana
  - University of Maryland, Baltimore, Maryland
  - University of Minnesota, Minneapolis, Minnesota
  - New York Presbyterian Hospital, Columbia University Med. Ctr., New York, New York
  - Cleveland Clinic, Cleveland, Ohio
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Baylor College of Medicine, Houston, Texas
  - Inova Fairfax Hospital, Falls Church, Virginia
- University of Toronto, Toronto, Ontario, Canada

REFERENCES:
- [Background] Burkart GJ, Smaldone GC, Eldon MA, Venkataramanan R, Dauber J, Zeevi A, McCurry K, McKaveney TP, Corcoran TE, Griffith BP, Iacono AT. Lung deposition and pharmacokinetics of cyclosporine after aerosolization in lung transplant patients. Pharm Res. 2003 Feb;20(2):252-6. doi: 10.1023/a:1022275222207. PMID 12636164
- [Background] Iacono AT, Smaldone GC, Keenan RJ, Diot P, Dauber JH, Zeevi A, Burckart GJ, Griffith BP. Dose-related reversal of acute lung rejection by aerosolized cyclosporine. Am J Respir Crit Care Med. 1997 May;155(5):1690-8. doi: 10.1164/ajrccm.155.5.9154878.
- [Background] Keenan RJ, Iacono A, Dauber JH, Zeevi A, Yousem SA, Ohori NP, Burckart GJ, Kawai A, Smaldone GC, Griffith BP. Treatment of refractory acute allograft rejection with aerosolized cyclosporine in lung transplant recipients. J Thorac Cardiovasc Surg. 1997 Feb;113(2):335-40; discussion 340-1. doi: 10.1016/S0022-5223(97)70331-3. PMID 9040628
- [Background] Iacono A, Dauber J, Keenan R, Spichty K, Cai J, Grgurich W, Burckart G, Smaldone G, Pham S, Ohori NP, Yousem S, Williams P, Griffith B, Zeevi A. Interleukin 6 and interferon-gamma gene expression in lung transplant recipients with refractory acute cellular rejection: implications for monitoring and inhibition by treatment with aerosolized cyclosporine. Transplantation. 1997 Jul 27;64(2):263-9. doi: 10.1097/00007890-199707270-00015. PMID 9256185
- [Background] Iacono AT, Johnson BA, Grgurich WF, Youssef JG, Corcoran TE, Seiler DA, Dauber JH, Smaldone GC, Zeevi A, Yousem SA, Fung JJ, Burckart GJ, McCurry KR, Griffith BP. A randomized trial of inhaled cyclosporine in lung-transplant recipients. N Engl J Med. 2006 Jan 12;354(2):141-50. doi: 10.1056/NEJMoa043204. PMID 16407509
- [Background] Iacono AT, Corcoran TE, Griffith BP, Grgurich WF, Smith DA, Zeevi A, Smaldone GC, McCurry KR, Johnson BA, Dauber JH. Aerosol cyclosporin therapy in lung transplant recipients with bronchiolitis obliterans. Eur Respir J. 2004 Mar;23(3):384-90. doi: 10.1183/09031936.04.00058504. PMID 15065826
- [Background] Iacono AT, Keenan RJ, Duncan SR, Smaldone GC, Dauber JH, Paradis IL, Ohori NP, Grgurich WF, Burckart GJ, Zeevi A, Delgado E, O'Riordan TG, Zendarsky MM, Yousem SA, Griffith BP. Aerosolized cyclosporine in lung recipients with refractory chronic rejection. Am J Respir Crit Care Med. 1996 Apr;153(4 Pt 1):1451-5. doi: 10.1164/ajrccm.153.4.8616581.
- [Derived] Corcoran TE, Niven R, Verret W, Dilly S, Johnson BA. Lung deposition and pharmacokinetics of nebulized cyclosporine in lung transplant patients. J Aerosol Med Pulm Drug Deliv. 2014 Jun;27(3):178-84. doi: 10.1089/jamp.2013.1042. Epub 2013 May 13. PMID 23668548